CLINICAL TRIAL: NCT00650676
Title: The Effect of Somatosensory Cue on Postural Stability in Blinded Persons
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Itshak Melzer PhD, PT, Ben-Gurion University of the Negev
Other Study IDs: sor464308ctil; MY4643
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A

SUMMARY:
Blind Adults that willing to participate in the study will be tested with well-established measuring techniques of Balance control using force plate in the movement and Rehabilitation Laboratory at Ben-Gurion University. An automated algorithm will be used to extract standardized stabilogram-diffusion parameters from each of the COP data sets collected during quiet standing. These parameters include diffusion coefficients, critical displacement, critical time and scaling exponents for both lateral and anterior-posterior sway directions (Collins & De Luca, 1993). the subjects will be tested in 3 task conditions (eyes blindfolded, eyes blindfolded holding stick, eyes blindfolded holding a dog). Participants will be required to stand on the platform 10 times for 30 s For each trial, they will be instructed to sway as little as possible.

ELIGIBILITY:
Inclusion Criteria:

* Blind persons
* Able to stand safely for 30 seconds
* Able to walk independently
* Hip OA prior THA

Exclusion Criteria:

* Stroke or other neurological diseases
* Orthopedic surgery at the past year

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 blind persons and 30 control
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
SDF parameters | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Itshak Melzer, PhD, Principal Investigator — Ben-gurion University of the Negev, Beer-Sheva, Israel; Ronit Yagev, MD, Study Chair — Soroka University Medical Centar
Locations (1):
- Soroka University Medical Center, Beersheba, Israel